CLINICAL TRIAL: NCT04855058
Title: Long Term Follow-Up of Traumatic Fracture Patients Treated With Integrated Complementary and Alternative Medicine: Observational Study
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2020-15
Record Dates: First submitted 2021-04-12; First posted 2021-04-22 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Fractures, Bone; Medicine, Korean Traditional
Keywords: acupuncture therapy; herbal medicine
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: online survey(or phone survey) — A questionnaire about the current symptoms and satisfaction for received treatment will be conducted over google survey(or the phone survey) for patients.

SUMMARY:
The purpose of this study is to reveal the effectiveness of integrative Korean medicine for trauma fracture by observation inpatients treated with integrative Korean medicine.

This study is a prospective observational study. The subjects for study are patients diagnosed with fracture and who have been admitted to five Jaseng Hospital of Korean medicine (Gangnam, Bucheon, Daejeon, Bundang and Haeundae) for 2017.03-2020.08.

Medical records of selected patients will be analyzed, and online google surveys(or telephone) will be conducted for each patient. The survey questions are Numeric rating scale (NRS), quality of life, and Patient Global Impression of Change (PGIC), etc.

ELIGIBILITY:
Inclusion Criteria:

1. 19-85 years old
2. Pateints who have been admitted to five Jaseng Hospital of Korean medicine (Gangnam, Bucheon, Daejeon, Bundang and Haeundae) and hospitalized 5 days or more
3. fracture caused by trauma
4. Patients have agreed to participate the study.

Exclusion Criteria:

1. pathological fracture, stress fracture
2. Open fracture
3. The cause of pain is due to other disease, not the fracture: tumors, fibromyalgia, rheumatoid arthritis, gout, etc.
4. Patients who are difficult to complete the research questionaire because of communication, mental or physical capabilities.
5. lack of data of collection
6. Patients deemed unable to participate in the clinical research by other researchers

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects for study are patients diagnosed with fracture and who have been admitted to five Jaseng Hospital of Korean medicine (Gangnam, Bucheon, Daejeon, Bundang and Haeundae) for 2017.03-2020.08.
Sampling Method: Non-Probability Sample
Enrollment: 665 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Numeric rating scale(NRS) to longterm f/u survey | baseline(admission), week 1, 2, 3, 4, 5, 6, 7, day of Discharge(up to week 8), finish f/u survey by June 2021
  NRS uses an 11-point scale to evaluate current neck pain and radiating pain where no pain is indicated by '0', and the worst pain imaginable by '10'.

SECONDARY OUTCOMES:
The five level version of EuroQol-5 Dimension (EQ-5D) | baseline(admission), week 2, 4, 6, day of Discharge(up to week 8), finish f/u survey by June 2021
  EQ-5D is most widely used as a method of indirectly calculating the quality of life from various aspects. The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about) In this study, the validated Korean version questionnaire will be used
Oswestry disability index (ODI) | baseline(admission), week 2, 4, 6, day of Discharge(up to week 8), finish f/u survey by June 2021
  The ODI is a 10-item questionnaire developed to evaluate the degree of disability for low back pain. Each item is divided into 6 levels, and 0 to 5 points are awarded. The higher the score, the greater the degree of disability. We will conduct an validated Korean ODI questionnaire(to L-SPINE, T-SPINE and sacrum fracture)
Neck Disability Index (NDI) | baseline(admission), week 2, 4, 6, day of Discharge(up to week 8), finish f/u survey by June 2021
  NDI is a 10-item questionnaire developed to evaluate the degree of disability for neck back pain. Each item is divided into 6 levels, and 0 to 5 points are awarded. The higher the score, the greater the degree of disability. We will conduct an validated Korean NDI questionnaire (to C-SPINE fracture)
Shoulder Pain and Disability Index (SPADI) | baseline(admission), week 2, 4, 6, day of Discharge(up to week 8), finish f/u survey by June 2021
  The Shoulder Pain and Disability Index (SPADI) is a patient completed questionnaire with 13 items assessing pain level and extent of difficulty with ADLs requiring the use of the upper extremities. The pain subscale has 5-items and the Disability subscale has 8-items. We will conduct an validated Korean SPADI questionnaire (to shoulder fracture)
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline(admission), week 2, 4, 6, day of Discharge(up to week 8), finish f/u survey by June 2021
  WOMAC is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). We will conduct an validated Korean WOMAC questionnaire. (to knee fracture)
Quick Disabilities of the Arm, Shoulder, and Hand questionnaire (QuickDASH) | at finish f/u survey by June 2021
  The DASH, an instrument that evaluates upper ex- tremity disabilities, has advantages for analyzing the overall function of the upper extremity. The 30 items in the questionnaire ask about different upper extremity disabilities in terms of symptoms, physical functions, social functions, and psychological problems. A shorter version of DASH, known as Quick Disabilities of the Arm, Shoulder, and Hand questionnaire (QuickDASH), consists of 11 items from the original DASH. We will conduct an validated Korean Quick DASH questionnaire. (to clavicle, arm and hand fracture)
the Hip Disability and Osteoarthritis Outcome Score(HOOS) | at finish f/u survey by June 2021
  HOOS is developed as an instrument to assess the patients' opinion about their hip and associated problems. HOOS consists of 5 subscales; Pain, other Symptoms, Function in dailyliving (ADL). Standardized answer options are given and each question gets a score from 0 to 4. A normalized score(100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The result can be plotted as an outcome profile. We will conduct an validated Korean HOOS questionnaire.(to hip joint , ilium, ischium, and pubis fracture)
the Foot Function Index (FFI) | at finish f/u survey by June 2021
  The FFI was developed to measure the effect of foot problems on function in terms of pain and disability. The FFI is a self-administered index consisting of 23 items divided into 3 scales(limitation, pain, and disability). Korean FFI questionnaire was validated in only 2 scales(pain, disability), and we use only pain scale of FFI (to ankle and foot fracture).
Symptoms of RIB,STERNUM fracture | at finish f/u survey by June 2021
  There is no validated worldwide used questionnaire. so we use 4 questions about symptoms associated with rib and sternum fracture, based on previous article. (pain during deep breathing, coughing, turning over the body, and sleeping)
Patient Global Impression of Change (PGIC) | at finish f/u survey by June 2021
  PGIC is an indicator that evaluates the improvement of patients in 7 steps, and the subject responds with improvement of functional limitation after treatment with 7 likert. (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse).
hanbangchilyo manjogdo (Satisfaction with integrative Korean medicine) | at finish f/u survey by June 2021
  5 answer options are given: very satisfied, a little satisfied, moderate, a little dissatisfied, very dissatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Jaseng Medical Foundation, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No